CLINICAL TRIAL: NCT07206316
Title: Health-economic Evaluation of the IPS (Individual Placement and Support) Model for Helping People With Severe Mental Disorders Access Employment in the Ordinary Labor Market, Compared to Standard Methods of Helping People Return to Work: a Prospective Real-life Study
Acronym: MEDECO-IPS
Status: Not yet recruiting | Type: Observational
Sponsor: University Hospital, Tours (Other)
Responsible Party: Sponsor
Other Study IDs: DR240280-MEDECO-IPS
Record Dates: First submitted 2025-09-25; First posted 2025-10-03 (Actual); Last update posted 2025-10-03 (Actual); Status verified 2025-09

CONDITIONS: Severe Mental Disorders
Keywords: Individual Placement and Support; Health-economic evaluation
MeSH Terms: conditions — Mental Disorders

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- IPS (Individual Placement and Support) practice model: patients benefiting from the IPS (Individual Placement and Support) practice model for assistance in accessing employment
  Interventions: Other: Individual Placement and Support Model
- standard method: patients benefiting from the standard method for assistance in accessing employment
  Interventions: Other: Standard Method

INTERVENTIONS:
Other: Individual Placement and Support Model — The Individual Placement and Support (IPS) model is an employment support program specifically designed for people with severe mental illness (Bond, Drake, & Becker, 2012). The core philosophy of IPS is that anyone can obtain competitive employment in the open labor market, provided it is the right job combined with appropriate support.
  IPS support is delivered by a job coach, specifically trained in this model, who devotes their entire working time to assisting patients in their vocational integration.
  Groups: IPS (Individual Placement and Support) practice model
Other: Standard Method — In psychiatric wards, patients who wish to do so are usually offered support to initiate the process of returning to competitive employment in the open labor market. This assistance is provided by the social workers (such as social workers or educators) within the care unit.
  Groups: standard method

SUMMARY:
The Individual Placement and Support (IPS) model was developed in the United States in the 1990s to help people with severe mental health issues get back into regular jobs. This model is based on the idea that a quick job search that takes into account what patients want, followed by ongoing and intensive support in the community, is especially good for this group. To date, although the effectiveness of the IPS model has been widely demonstrated (for a review, see Metcalfe et al., 2018), only a few studies have evaluated its efficiency in foreign contexts (Knapp et al., 2013; Christensen et al., 2020).

Although the IPS model has been in place in France for around ten years, no studies have yet been conducted to validate its efficiency in the French healthcare system.

The main objective of this prospective, real-life, multicenter study is to evaluate the efficiency of the IPS practice model compared to the conventional method of follow-up by social workers for patients with severe mental illness in terms of cost per additional day worked, from a collective perspective.

ELIGIBILITY:
Inclusion Criteria:

* Aged ≥ 18 years
* Participant with a chronic psychiatric disorder causing significant functional impairment
* Unemployed
* Wishing to return to competitive employment in the open labor market
* Informed about the study and consenting to participate
* Able to read french

Exclusion Criteria:

* Individuals not eligible for legal employment due to irregular residency status in France
* Individuals not affiliated with a social security system
* Individuals wishing to work in a sheltered/protected setting
* Individuals currently enrolled in a training program
* Individuals refusing to participate in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients with severe mental disorders treated in adult psychiatric wards and receiving support to return to competitive employment in the open labor market in France
Sampling Method: Non-Probability Sample
Enrollment: 234 (Estimated)
Dates: Start 2025-10-02 (Estimated); Primary Completion 2030-03 (Estimated); Study Completion 2030-03 (Estimated)

PRIMARY OUTCOMES:
Efficiency of the IPS practice model compared to the conventional method of follow-up by social workers for patients with severe mental illness | 18 months
  Incremental cost-effectiveness ratio (ICER) expressed as cost per additional day worked at 18 months, from a collective perspective, of the IPS practice model in patients with severe mental disorders.

SECONDARY OUTCOMES:
Efficiency of the IPS model compared to the conventional method of monitoring by social workers among patients with severe mental illness | 18 months
  Incremental cost-utility ratio (ICUR) expressed as "cost/QALY gained at 18 months, from a collective perspective, of the IPS model in patients with severe mental disorders.
Cost-benefit ratio of the IPS practice model compared to the conventional method of follow-up by social workers for patients with severe mental illness, | 18 months
  Benefit-cost ratio of the IPS model compared to the conventional method of follow-up by social workers at 18 months, from a societal perspective, among patients with severe mental illness
Budgetary impact on the French national health insurance system (AM) of changes in clinical practices with regard to the two types of support for returning to work. | 5 years
  Budgetary impact for the Health Insurance system per year and over 5 years of the evolution of practices with regard to the two types of support for return to work
Compare work productivity and activity disorders between the two groups. | 0, 6, 12 and 18 months
  Comparison of scores on the questionnaire on work productivity and activity impairment (French version of the Work Productivity and Activity Impairment, WPAI)
Compare the rate of hospital care use between the two groups. | 18 months
  Comparison of the number of hospitalizations, number of visits to psychiatric emergency rooms, and number of day hospital visits between the two groups
Impact of a return to work on patients' level of recovery and overall health. | 18 months
  Comparison of scores on a clinical scale of recovery and overall health (French version of the Recovery Assessment Scale, RAS) between the two groups
Impact of a return to work on patients' level of social cognition. | 18 months
  Comparison of scores on the ACSo clinical social cognition scale between the two groups
Impact of a return to work on patients' cognitive functioning | 18 months
  Comparison of scores on the clinical cognitive functioning scale (French version of the Subjective Scale to Investigate Cognition in Schizophrenia, SSTICS) between the two groups

CONTACTS AND LOCATIONS:
Locations (11):
- France (11):
  - CH Cesame, Angers
  - CH George Sand, Bourges
  - Centre hospitalier Le Vinatier, Bron
  - CHI EPSM Oise, Clermont
  - University hospital, Clermont-Ferrand
  - Centre Hospitalier Marius Lacroix, La Rochelle
  - CH Esquirol, Limoges
  - Hôpital la Colombière, Montpellier
  - PRISM 45, Orléans
  - CH Le Rouvray, Rouen
  - University hospital, Tours

IPD SHARING:
Plan to Share IPD: Undecided